CLINICAL TRIAL: NCT00000290
Title: Stress Hormones and Human Cocaine Use
Brief Title: Stress Hormones and Human Cocaine Use - 7
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Minnesota (Other)
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09259-7; P50-09259-7
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Cocaine

INTERVENTIONS:
Drug: Cocaine

SUMMARY:
The purpose of this study is to determine the HPA axis and adrenergic system activation in response to cocaine administration.

DETAILED DESCRIPTION:
The goal of this study was to investigate the role of sympathetic-adrenal medullary (SAM) and hy0pothalamo-pituitary-adrenal (HPA) systems in mediating the addictive effects of cocaine. A toal of 6 male subjects were enrolled for this 5 day inpatient study. Subjects were assigned to either cocaine (32mg /70kg iv) or placebo (saline iv) treatment during the first experimental sessions and were crossed over to the alternative treatment during the second experimental session. Endpoints that were followed during the experimental sessions included neuroendocrine (serum epinephrine, norepinephrine and cortisol levels), physological (heart rate/blood pressure, EKG) and subjective measures (Beck Depression Inventory, Craving Questionnaire). We hypothesized that cocaine administration would lead to increased blood levels of norpinephrine, epinephrine and cortisol in cocaine dependent subjects.

ELIGIBILITY:
Inclusion Criteria:

Males between the ages of 20-45. History of smoked or intravenous cocaine use on the average of at least once a week over a 6 month period. Current history of good health and normal EKG.

Exclusion Criteria:

History of suicide attempt, bipolar disorder, schizophrenia, or generalized anxiety disorder. Current problem with major depressive disorder. Current use of alcohol or other drugs on a daily basis. History of major medical illnesses. Currently on parole, probation or a legal history of violence. Treatment for chemical dependency within the past 6 months. History of sensitivity to tricyclic compounds or other prescription drugs. Use of any psychotropic drugs including MAOIs in the past 6 months.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1997-05; Study Completion 2001-12

PRIMARY OUTCOMES:
Physiological measures
Biochemical

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Presented at CPDD, 6/13/99. None